CLINICAL TRIAL: NCT05606757
Title: A Phase 2b Double-Blind, Placebo-Controlled, Adaptive, Dose-Escalation Study to Evaluate the Safety and Efficacy of OnabotulinumtoxinA for the Achievement of Primary Fascial Closure Without the Use of Component Separation Technique, in Subjects Undergoing Open Abdominal Ventral Hernia Repair
Brief Title: A Study to Evaluate Adverse Events and Effectiveness of OnabotulinumtoxinA in Participants Undergoing Open Abdominal Ventral Hernia Repair for the Achievement of Primary Fascial Closure Without the Use of Component Separation Technique
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-779
Record Dates: First submitted 2022-11-01; First posted 2022-11-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Ventral Hernia; Abdominal Hernia
Keywords: OnabotulinumtoxinA; BOTOX; Abdomen; Primary fascial closure
MeSH Terms: conditions — Hernia, Ventral; Hernia, Abdominal | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Cohort 1, BOTOX Dose A (Experimental): Participants will receive BOTOX Dose A
  Interventions: Drug: BOTOX Dose A
- Cohort 1, BOTOX Dose B (Experimental): Participants will receive BOTOX Dose B.
  Interventions: Drug: BOTOX Dose B
- Cohort 1, Placebo (Placebo Comparator): Participants will receive placebo for BOTOX.
  Interventions: Drug: Placebo for BOTOX
- Cohort 2, BOTOX Dose A (Experimental): Participants will receive BOTOX Dose A
  Interventions: Drug: BOTOX Dose A
- Cohort 2, BOTOX Dose B (Experimental): Participants will receive BOTOX Dose B
  Interventions: Drug: BOTOX Dose B
- Cohort 2, BOTOX Dose C (Experimental): Participants will receive BOTOX Dose C
  Interventions: Drug: BOTOX Dose C
- Cohort 2, Placebo (Placebo Comparator): Participants will receive placebo for BOTOX
  Interventions: Drug: Placebo for BOTOX
- Cohort 3, BOTOX Dose A (Experimental): Participants will receive BOTOX Dose A
  Interventions: Drug: BOTOX Dose A
- Cohort 3, BOTOX Dose B (Experimental): Participants will receive BOTOX Dose B.
  Interventions: Drug: BOTOX Dose B
- Cohort 3, BOTOX Dose C (Experimental): Participants will receive BOTOX Dose C.
  Interventions: Drug: BOTOX Dose C
- Cohort 3, Placebo (Experimental): Participants will receive placebo for BOTOX.
  Interventions: Drug: Placebo for BOTOX

INTERVENTIONS:
Drug: BOTOX Dose A — Injection; intramuscular
  Other Names: OnabotulinumtoxinA
  Arms: Cohort 1, BOTOX Dose A; Cohort 2, BOTOX Dose A; Cohort 3, BOTOX Dose A
Drug: Placebo for BOTOX — Placebo
  Arms: Cohort 1, Placebo; Cohort 2, Placebo; Cohort 3, Placebo
Drug: BOTOX Dose B — Injection; intramuscular
  Other Names: OnabotulinumtoxinA
  Arms: Cohort 1, BOTOX Dose B; Cohort 2, BOTOX Dose B; Cohort 3, BOTOX Dose B
Drug: BOTOX Dose C — Injection; intramuscular
  Other Names: OnabotulinumtoxinA
  Arms: Cohort 2, BOTOX Dose C; Cohort 3, BOTOX Dose C

SUMMARY:
Ventral hernias form when there is a loss of integrity of the abdominal wall muscles. Abdominal hernias can expand and can cause severe pain as the abdominal wall weakens. The purpose of this study is to evaluate the safety and efficacy of a range of onabotulinumtoxinA (BOTOX) doses to achieve primary fascial closure (PFC) without use of component separation technique (CST) in ventral hernia surgical repair.

BOTOX is an investigational drug being developed for the treatment of ventral hernias. In this dose escalation study, participants will be placed in 1 of 3 cohorts. Cohort 1 will be randomized to receive placebo or 1 of 2 BOTOX doses, after which time Cohort 2 will be randomized to receive placebo or 1 of 3 BOTOX doses. Participants in Cohort 3 will be randomized to receive placebo or 1 of 3 BOTOX doses. Adult participants undergoing open abdominal ventral hernia repair will be enrolled. Around 200 participants will be enrolled in the study at approximately 20 sites in the United States.

Participants will receive a single intramuscular injection of BOTOX Dose A, BOTOX Dose B, BOTOX Dose C, or placebo.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will be followed for approximately 3 months after surgery and will receive a follow-up phone call 30 days (+/-) their last study visit. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant is in good health as determined by medical history, vital signs, and investigator's judgment, including no known active pandemic infection.
* Body Mass Index (BMI) at screening is <= 40 kg/m2.
* Participant meets the following disease activity criteria:

  * Intact abdominal wall muscles (defined as no prior dissection to the lateral abdominal wall complex) based on screening CT scan.
  * Midline ventral hernia requiring surgical repair, at least 6 cm, and not more than 18 cm in transverse defect width at the widest part of the of the hernia defect, as assessed on CT scan by the investigator.
  * Any portion of the ventral hernia does not extend > 3 cm into the M1 subxiphoid zone or into the M5 zone using the 2009 classification by the European Hernia Society.
  * No history of prior onlay hernia mesh wider than rectus.
  * No hernia with loss of domain >20% as determined by the investigator, using Sabbagh method.

Exclusion Criteria:

* Presence of a medical condition that may put the participant at increased risk with exposure to onabotulinumtoxinA, including diagnosed muscular dystrophy (e.g., Duchenne's muscular dystrophy), myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, mitochondrial disease, or any other significant disease which might interfere with neuromuscular function.
* Presence or history of any of the following within 3 months prior to the randomization visit that may indicate a vulnerable respiratory state per the investigator's clinical judgment, for example, aspiration pneumonia, lower respiratory tract infections, uncontrolled asthma, severe chronic obstructive pulmonary disease, or otherwise compromised respiratory function.
* History of ongoing or anticipated need to perform progressive preoperative pneumoperitoneum or other tissue expansion technique for repair of ventral hernia.
* Planned ostomy reversal, panniculectomy bariatric procedure, or vascular procedure requiring anticoagulants during the study.
* History of abdominal or hernia repair surgery requiring hospitalization within 6 months prior to screening.
* History of a contraindication to BOTOX and/or hypersensitivity reactions to BOTOX.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-07 (Estimated); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with achievement of primary fascial closure (PFC) without the use of component separation techniques (CST) in open ventral hernia surgical repair | Up to 4 Months
  PFC will be defined as the ability to achieve fascia to fascia midline approximation. CST will be defined as the release of the external oblique muscle or the transection of transversus abdominis muscle (known as posterior component separation with transversus abdominis release (TAR).

SECONDARY OUTCOMES:
Percentage of participants with achievement of PFC | Up to 4 Months
  PFC will be defined as the ability to achieve fascia to fascia midline approximation.
Percentage of participants with usage of CST for the purpose of PFC | Up to 4 Months
  CST will be defined as the release of the external oblique muscle or the transection of transversus abdominis muscle (known as posterior component separation with transversus abdominis release (TAR).
Number of lateral abdominal wall muscles released among participants who required CST use to achieve PFC as reported by the operating surgeon | Up to 4 Months
  Lateral abdominal wall muscles are released by TAR and external oblique release (unilateral or bilateral)
Change in length of lateral abdominal wall complex | Up to 4 Months
  Change in length of lateral abdominal wall complex as measured by abdominal CT scan in supine position prior to surgical repair will be assessed.
Change in Width to the Hernia Defect | Up to 4 Months
  Change from screening in width to the hernia defect as measured by abdominal CT scan in supine position prior to surgical repair will be assessed.
Change from screening in length of lateral abdominal wall complex | Up to 4 Months
  Change from screening in length of lateral abdominal wall complex as measured by abdominal CT scan performing Valsalva maneuver prior to surgical repair will be assessed.
Change from screening in width to the hernia defect | Up to 4 Months
  Change from screening in width to the hernia defect as measured by abdominal CT scan performing Valsalva maneuver prior to surgical repair

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - NYU Langone Hospital - Long Island /ID# 251280, Mineola, New York
  - Atrium Health Carolinas Medical Center /ID# 247711, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/